CLINICAL TRIAL: NCT04042766
Title: Laser Vaginal Treatment for GSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Innovation Fund of the Alternative Funding Plan from the Academic Health Sciences Centres of Ontario (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 094-2019
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-04

CONDITIONS: Menopausal Urethral Atrophy; Vulvar Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser treatment (Active Comparator)
  Interventions: Procedure: laser vaginal treatment
- sham treatment (Sham Comparator)
  Interventions: Procedure: laser vaginal treatment

INTERVENTIONS:
Procedure: laser vaginal treatment — Er:YAG laser

SUMMARY:
Genitourinary Syndrome of Menopause (GSM) due to low estrogen levels affects about half of post-menopausal women and may have a dramatic impact on women's quality of life. Women complain of vaginal dryness, itching, discomfort, malodour, painful intercourse and may have urinary urgency, irritation, bladder/urethral pain and recurring bladder infections. First-line therapies include vaginal moisturizers, lubricants and estrogen (either oral or with vaginal cream/tablets). While these therapies are effective, the ongoing costs and the resistance to the indefinite use of vaginal creams/inserts is a challenge to the continued use of these therapies. Recently, an innovative laser therapy has been used to treat women with GSM. A randomized controlled trial (RCT) to study how effective the laser is to treat women with GSM is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 45-70 years;
2. 2 or more years since last natural menstrual period, or surgical menopause (bilateral oophorectomy);
3. at least 1 vaginal symptom reported from the following list, experienced for the past 30 days which is moderate or severe at least once a week: dryness | itching | irritation | soreness/pain | dyspareunia;
4. no concurrent or new planned treatment for GSM during the treatment period and the 3 months following it;
5. vaginal anatomy allows for laser therapy; 6) willing and able to comply with the study protocol.

Exclusion Criteria:

1. Patient is pregnant/lactating
2. unexplained abnormal genital bleeding
3. current acute vaginal/ bladder infection
4. antibiotic use the past 30 days;
5. women under age 55 with endometrial ablation/ hysterectomy/ at least one ovary;
6. concurrent use of any other new GSM treatment
7. pelvic surgery <3 months
8. current treatment for chronic pelvic pain

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
subjective measure of change in: the patient's most bothersome symptom | Baseline and 3 months after treatment start
  The most bothersome symptom of GSM (vaginal dryness, discomfort, itching, dyspareunia, urinary urgency, dysuria) will be identified and its severity rated on a standardized 4-point scale: 0=none, 1=mild, 2=moderate, 3=severe

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lee, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No